CLINICAL TRIAL: NCT00120614
Title: Improving Outcomes of LBW Premature Infants and Parents
Brief Title: Educational/Behavioral Intervention Program for Parents of Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 06990; 5RO1MR5077-5
Record Dates: First submitted 2005-07-07; First posted 2005-07-18 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Premature Birth
Keywords: Premature Infant; Premature Birth; Parenting Interventions; NICU Interventional studies; Parental coping; Low birthweight infant; Coping Behavior; Infant, Premature
MeSH Terms: conditions — Premature Birth

INTERVENTIONS:
Behavioral: Premature infant behavior and development information
Behavioral: Parental activities to support premature infant information

SUMMARY:
The purpose of this study is to determine whether beginning an enriched educational/behavioral program for parents of premature infants, very early in the Neonatal Intensive Care Unit (NICU) stay, and lasting until the child is 3 years old, has beneficial results for both the parents and their infants.

The hospital phase of the program gives parents an understanding of what to expect in the NICU environment; physical characteristics and needs of their premature baby; and how and when to best support their infant's development during this time. The information given during the home phase of the program continues with information specific to the growth and development and the effective parenting of an infant/toddler who has been born prematurely.

It is believed that this information will help decrease parents' stress, anxiety and depression levels that can be related to giving birth to a premature infant. It is also expected that it will strengthen the mother's and father's ability to parent their premature child in a way that will help support their child's brain development and learning ability and to also decrease negative behaviors as the child grows.

DETAILED DESCRIPTION:
The incidence of premature and low birthweight (LBW) births continues to climb in the U.S. despite increased efforts to prevent it. Interventions to enhance coping in parents of infants in an attempt to improve both parent and child outcomes have not kept pace with the rapid technological advances to sustain survival for these medically compromised infants. Consequently, there is an urgent need to develop and evaluate coping interventions for parents of LBW premature infants in order to facilitate effective clinical practice strategies that are empirically based.

The primary objective for this study is to evaluate the short- and long-term effects of a theoretically-driven intervention program (COPE: Creating Opportunities for Parent Empowerment) on the process and outcomes of mothers and fathers/significant others' (SOs) coping with a LBW premature infant and infant developmental outcomes. The secondary objectives are to:

* Explore how the coping process and outcomes of mothers and fathers/significant others together contribute to the outcomes of LBW premature infants;
* Determine the cost-effectiveness of the COPE program; and
* Explore what factors moderate the effects of the intervention (e.g., family structure, SES, birthweight, disability, and infant temperament).

In this randomized clinical trial, the investigators are testing the following hypotheses separately for mothers and for fathers/significant others:

* Mothers/fathers who receive the COPE program will report less anxiety, depression, and stress related to the NICU environment than mothers/fathers who receive the comparison program;
* Mothers/fathers who receive the COPE program will demonstrate a higher quality of parenting during hospitalization than mothers/fathers who receive the comparison program;
* Mothers/fathers who receive the COPE program will report less anxiety and depression following hospitalization than mothers/fathers who receive the comparison program;
* Mothers/fathers who receive the COPE program will perceive their children as less vulnerable than mothers/fathers who receive the comparison program;
* Fathers who receive the COPE program will report greater involvement in their infants' lives (average time spent with infant per week) than fathers who receive the comparison program;
* Infants of mothers/fathers who receive the COPE program will have greater cognitive development than infants of mothers/fathers in the comparison program;
* Children of mothers/fathers in the COPE program will have less negative behaviors at 2 years corrected age than children of mothers/fathers in the comparison program;
* The proposed model to explain the effects of the COPE program on the process and outcomes of parental coping and infant outcomes will be supported for mothers and for fathers.

In addition, the following study questions will be answered:

* How do parental beliefs and coping outcomes of both mothers and fathers together contribute to the outcomes of LBW premature infants?
* Are there reciprocal effects between parent and child outcomes as well as parental emotional and functional coping outcomes?
* How do infant cognitive development and parental coping outcomes change over time within the subjects and between the experimental groups?
* What factors moderate the effects of the intervention on child outcomes (e.g., family structure, SES, birth-weight, disability, and infant temperament)?
* What is the incremental cost of the COPE intervention compared to the comparison group, when the health care sector perspective is considered?
* What is the incremental cost of the COPE intervention compared to the comparison group intervention, when the societal perspective is considered?
* How sensitive are the findings in these economic evaluations to the assumptions and parameter estimates made in the analyses?

The first 3 years of life and the quality of early parent-child relations are principal building blocks for adult cognitive and emotional functioning. However, investigators have found that parents have impaired relationships with their premature infants, providing heightened stimulation to the infants at inappropriate times in hopes of increasing responsiveness to them. These dysfunctional patterns place parents at risk for negative emotions and parenting outcomes and place children at risk for emotional, behavioral, and developmental problems. Therefore, early interventions are critical to decrease the negative effects of prematurity on parenting and parent-infant interactions. Early intervention may be a critical key to future successful programs with parents and their premature infants because it is recognized that, once a trajectory of parent-infant interaction is initiated, changes are difficult to implement and even harder to sustain; this program has the potential to benefit a significant number of LBW premature infants and their parents across the country.

A randomized block design with repeated measures is being used. Subjects at each of two study sites are randomly assigned to the COPE or comparison group by 4-week periods of time. Using random assignment at each site will allow for assessment of an interaction effect as part of the data analytic strategy. Based on the average NICU stay in the pilot study (mean = 29.6 days), the decision to use 4-week blocks of time was made to decrease the likelihood of parent to parent and staff to parent contamination which would be more likely with individual randomization.

The COPE program provides parents with: (a) information on the appearance and behavioral characteristics of premature infants and information on how parents can participate in their infant's care, meet their infant's needs, enhance the quality of interaction with their infant, and facilitate their infant's development (parental role information); and (b) activities that assist parents in implementing the experimental information. The content of the COPE program is driven by the theoretical framework, developmental theory, the literature review, interventions found to be effective in previous studies, and prior work by the research team.

The COPE program consists of 7 phases. Phase I (within 2 to 4 days after the infant's NICU admission) consists of audiotaped information. A written copy of the information is also provided for parents to read as they listen to the audiotape. Also, parents are given their first set of parenting activities that consist of: (a) identifying the special characteristics of their baby; and (b) keeping a record of milestones that their baby achieves while in the NICU. Phase II (within 2 to 4 days after the first intervention) consists of audiotaped and written information that reinforce the critical content of the initial audiotape and provides supplemental information on: (a) premature infants' behaviors and development; and (b) further suggestions regarding how parents can participate in their infant's care and enhance their infant's development. Additional activities are introduced to parents that consist of: (a) identifying the special characteristics of their baby at this time; and (b) recognizing their baby's stress cues as well as cues that signal readiness for communication. The parent activities are designed to: (a) supplement mothers and fathers' existing parenting repertoire by providing them with parent activities specific to the situation; (b) increase parents' confidence and certainty regarding how they can best meet their infant's needs; and (c) enhance infant developmental outcomes. Phase III (1 to 4 days prior to the infant's discharge to home) consists of developmentally appropriate information, including specific details about infant states and the best times for mothers and fathers to interact with their infant. The audiotape also contains parental role information regarding how to smooth the transition from hospital to home as well as how to continue to foster a positive mother/father-baby relationship. Parent activities during Phase III include: (a) continuing to assist parents in recognizing their baby's cues; and (b) helping parents to recognize strategies that help their baby when he or she is stressed. The Phase III intervention was planned for this window of time because discharge to home is empirically supported as a stressful transition for parents.

Phase IV (within 1 week after discharge) is delivered in the parents' home. Audiotaped information at this time contains information specific to continued growth and development of the infant and suggestions for fostering a positive parent-infant relationship. Further parenting activities are given to mothers and fathers that outline specific things for them to do with their infant to foster his or her cognitive development (e.g. age appropriate games and songs). One of these activities is a book, The Little Engine that Could, for parents to read to their infants. Emphasis is placed upon interacting when the infant is most receptive to stimuli (e.g., while in the quiet alert state). Phase V (2 months corrected age) is also delivered in the parents' home. Parents again receive audiotaped and written information about appropriate upcoming developmental milestones and how they can enhance their infant's development. Emphasis is placed on specific age-appropriate information about: (a) their infant's developmental characteristics; (b) typical sleep, crying, and temperament patterns; and (c) strategies to foster their infant's cognitive and social development. The COPE information places emphasis on assessing their infants based on their corrected versus chronological age. Parenting activities in this phase of the intervention include: (a) rattle play; (b) playing "peek-a-boo"; (c) repeating an action; (d) tasting and touching to explore; and (e) vocalizing to take a turn. At Phase VI (9 months corrected age) parents are provided with audiotaped information that: (a) educates them regarding what to expect in their infant's upcoming development; and (b) provides suggestions for enhancing their child's development. Because mothers of LBW premature infants frequently continue to view their children as "fragile" through the preschool years and engage in overprotective parenting, this intervention focuses on the importance of letting toddlers engage in autonomy, exploration, self-initiation, and self-assertion. The COPE information outlines parenting strategies that foster positive attributes in the children in addition to teaching age-appropriate limits. Parenting activities to enhance development in this phase include: (a) learning the meaning of "no"; (b) learning about colors and sizes; (c) finger-painting; (d) reading; and (e) identifying body parts. Phase VII (18 months corrected age) information continues to emphasize the importance of allowing the child to develop autonomy, self-initiation, and appropriate exploration. Detailed information about the adverse effects of overprotective parenting is provided. Parents are given more information about how to engage in appropriate limit setting and discipline as well as strategies to continue to foster cognitive and social development with their toddler. The following parent-child activities are provided: (a) playdough and paint-recipes for fun; (b) matching objects to pictures; (c) learning to sort; (d) remembering where things belong; (e) learning to imitate two word phrases; and (f) recognizing and naming pictures.

The comparison program also consists of a series of audiotapes delivered at the same times as the 7 phases of the COPE program. Phases I and II audiotaped and written information contains information about the hospital services. The Phase III audiotape contains discharge information that is given to all parents. The audiotape provided during the Phase IV intervention contains information regarding immunizations. Phases V to VII audiotaped and written interventions focus on age appropriate child safety and nutrition issues.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 26 to 34 weeks inclusive
* Birthweight of less than 2500 grams
* Singleton birth
* Anticipated survival
* Not small for gestational age
* No severe handicapping conditions
* No Grade III or IV intraventricular hemorrhage
* Speaks and reads English

Exclusion Criteria:

* Parent/infant has positive drug testing
* Live outside of a 60 mile radius
* Had previous infants in a NICU
* Significant mental health history

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 260
Dates: Start 2001-09; Study Completion 2007-06

PRIMARY OUTCOMES:
Measures of emotional coping (mother/father/SO): State Anxiety Inventory: Phase I through VII Interventions and Observations (with exception of Phase II Observation)
Beck Depression Inventory II: Phase I through VII Interventions and Observations (with exception of Phase II Observation)
Parental stress related to NICU: Phase II (Intervention), Post hospital stress: Phase V, VI and VII (Intervention)
Infant/child outcomes: Infant cognitive development assessment: 6, 12, 24 months corrected age (Observation), Child behavior questionnaire: Phase VII (Observation)
Functional coping (mother/father/SO): Quality of parenting in the NICU: Phase II (Observation)
Quality of parenting at home: Phase VI (Observation), Parental problem solving: Phase V (Intervention and Observation)
Perception of child vulnerability: Phase VI and VII (Observation)
Parental/SO beliefs (Proposed Mediator): Parental Beliefs Scale questionnaire: Phase II and III (Intervention)

SECONDARY OUTCOMES:
Infant temperament (Proposed Moderator): Infant Temperament Questionnaires: Phase V, VI, VII (Intervention)
Cost outcomes (direct and indirect health care costs): Resource Utilization Questionnaire: 6, 12, 24 months corrected age (Observations)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Melnyk, PhD, RNC, Principal Investigator — Arizona State University/University of Rochester
Locations (2):
- United States (2):
  - University of Rochester Medical Center Neonatal Intensive Care Unit, Rochester, New York
  - Crouse Hospital, Syracuse, New York

REFERENCES:
- [Background] Melnyk BM, Alpert-Gillis L, Feinstein NF, Fairbanks E, Schultz-Czarniak J, Hust D, Sherman L, LeMoine C, Moldenhauer Z, Small L, Bender N, Sinkin RA. Improving cognitive development of low-birth-weight premature infants with the COPE program: a pilot study of the benefit of early NICU intervention with mothers. Res Nurs Health. 2001 Oct;24(5):373-89. doi: 10.1002/nur.1038. PMID 11746067
- [Background] Melnyk BM, Alpert-Gillis L, Feinstein NF, Crean HF, Johnson J, Fairbanks E, Small L, Rubenstein J, Slota M, Corbo-Richert B. Creating opportunities for parent empowerment: program effects on the mental health/coping outcomes of critically ill young children and their mothers. Pediatrics. 2004 Jun;113(6):e597-607. doi: 10.1542/peds.113.6.e597. PMID 15173543
- [Background] Melnyk BM, Feinstein NF, Fairbanks E. Effectiveness of informational/behavioral interventions with parents of low birth weight (LBW) premature infants: an evidence base to guide clinical practice. Pediatr Nurs. 2002 Sep-Oct;28(5):511-6. No abstract available. PMID 12424989